CLINICAL TRIAL: NCT06339515
Title: Design, Implementation and Evaluation of School Health Nursing Course Curriculum Based on Universal Design Model
Brief Title: Teaching School Health Nursing Course With Universal Design Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DuzceU-SBF-NYS-02
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2024-05

CONDITIONS: Nursing Education
MeSH Terms: interventions — Research Design

STUDY DESIGN:
Intervention Model Description: Universal Design Model for Learning
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- The research is a mixed method including quantitative and qualitative. (Other): Quantitative part of the research;Experimental:
  The curriculum, which will be prepared with the principles of the universal design model, will be implemented for 10 weeks, 3 lesson hours a weeks.
  The data of pre-invention study will be collected. Descriptive Characteristics Form, Critical Thinking Disposition Scale,Communication Skills Scale, Healthy Living Awareness Scale.
  Post-intervention data will be collected with Critical Thinking Disposition Scale,Communication Skills Scale, Healthy Living Awareness Scale.
  Qualitative part of the research:
  Experiences of Nursing Students: Student opinions will be taken weekly (Learning Diary) to determine the experiences of the students during the implementation process and at the end of the implementation.
  Reflective Diary: At the end of each session, the teacher will make a self-evaluation of the session.
  Interventions: Behavioral: Universal Design Model

INTERVENTIONS:
Behavioral: Universal Design Model — Universal design-based learning is based on the application of universal design approach principles to education. Universal design-based learning considers three broad networks of the brain to enable learning. These are recognition networks, strategic networks and affective networks. Universal design-based learning is a student-centered approach and curricula are designed to appeal to all students. Curricula consist of objectives, teaching methods, teaching materials and assessment and evaluation elements. Students' interests, needs and abilities are taken into consideration when designing curricula. Students' learning disabilities are identified and alternative practices are planned to eliminate these disabilities. All students are given equal opportunity to learn
  Other Names: Design, Implementation and Evaluation of School Health Nursing Course Curriculum Based on Universal Design Model

SUMMARY:
The aim of this study is to design, implement and evaluate the School Health Nursing course in the undergraduate nursing program using the universal design model.

DETAILED DESCRIPTION:
Nursing education has adopted technology, evidence-based practice, critical thinking, and collaborative work. In order for teaching to be successful, students with different characteristics should be addressed and diversity and flexibility should be taken into consideration in the teaching plan. In this context, the application of the principles of Universal Design for Learning (UDL) is recognized as an inclusive learning approach that can meet the diverse needs of nursing students. Despite this, UDL is not well known in nursing education. Nursing students are diverse in culture, abilities and challenges. IET is a logical and social model that supports a variety of learning modalities. Accessibility tools help to measure the effectiveness of faculty efforts to make nursing courses accessible to all. In a study conducted in the USA, 100 courses were analyzed 1 year apart for the use of accessibility software to measure faculty development and student participation in nursing courses over 2 academic terms (spring 2021 and 2022). It was found that course accessibility scores and student utilization increased significantly with SET. In a study designed in Canada for Covid-19 in the fall semester of 2020 using online IET-based teaching strategies, the undergraduate course given in the first year of nursing was evaluated with convergent mixed methods analysis. In the technology-enhanced face-to-face health sciences course where the principles of KET were applied, students were provided with a variety of means of representation, participation and expression. Students reported that the delivery of the course with SLT resulted in increased flexibility, socialization, reduced stress and increased achievement, and that they felt more empowered to make personal choices to best support their own learning. Given the relative ease of applying the principles of SLT to courses, it is thought that it can be easily integrated into nursing education.

Purpose: The aim of this study is to design, implement and evaluate the School Health Nursing course in the undergraduate nursing program using the universal design model.

Method: In the research, simultaneous mixed method will be used in which one-group pretest-posttest quasi-experimental model and qualitative research methods will be used together. The sample was found 27 with the "G. Power-3.1.9.2" program with a medium effect level (d=0.5), 5% margin of error (α=0.05) and 80% power (1β=0.80).

Data accumulation methods: Data, Descriptive Characteristics Form, Critical Thinking Disposition Scale,Communication Skills Scale, Healthy Living Awareness Scale, Experiences of Nursing Students Form (Learning Diary), Reflective Diary will be collected.

Relevant statistical techniques will be used to analyze quantitative data and content analysis method will be used to analyze qualitative data.

The curriculum, which will be prepared with the principles of the universal design model, will be implemented for 10 weeks, 3 lesson hours a weeks.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study

Exclusion Criteria:

* Students who decline to participate in the study
* Students who will not be able to participate in the application continuously

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
Critical Thinking Disposition Scale | Up to 10 weeks
  The scale was developed by Semerci in 2000. The scale consists of 49 items with 5 dimensions. Sub-themes of the scale are metacognition, flexibility, systematicity, tenacity-patience and open-mindedness. 14 of the items are in metacognition, 11 of these are in flexibility, 11 of these are in tenacitypatience, 8 of these are in open-mindedness. The Cronbach Alpha coefficient of the CDTH is 0.96. The maximum score that can be obtained from the scale is 245 and the minimum score is 49. the higher the total score, the higher the critical thinking.
Communication Skills Scale | Up to 10 weeks
  Communication skills scale helps to determine the communication skills of the students. Communication skills scale items centered on the factors of "competence", "discouragement", "body language" and "dignification" factors and there were 36 items in total. Cronbach's alpha coefficient of the scale is 0.89. The lowest score that can be obtained from the whole scale is 36 and the highest score is 180. In the sub-dimensions of the scale, the lowest score that can be obtained from the competence dimension is 12, the highest score is 60; the lowest score that can be obtained from the obstacle dimension is 13, the highest score is 65; the lowest score that can be obtained from the body language dimension is 5, the highest score is 25; the lowest score that can be obtained from the valuing dimension is 6, the highest score is 30 points. It can be concluded that the higher the scores obtained from the scale, the higher the level of communication skills.
Healthy Living Awareness | Up to 10 weeks
  Developed by Elif Özer, Necla Yılmaz in 2020, it has "Socialization", "Change", "Responsibility" and "Nutrition" sub-dimensions. It consists of 15 items. Cronbach's alpha coefficient of the scale is 0.81.The lowest score to be obtained from the scale is 15 and the highest score is 75. A high score on the scale is considered to indicate a high level of healthy life awareness.

CONTACTS AND LOCATIONS:
Overall Officials: Fahriye Hayırsever, PhD, Principal Investigator — Duzce University
Locations (1):
- Nuriye Yıldırım, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No